CLINICAL TRIAL: NCT00743808
Title: Improving Hypertension Control in Individuals With Diabetes
Brief Title: Hypertension and Diabetes Initiative - Improving Hypertension Control in Individuals With Diabetes
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Advocate Medical Group (Other); Baystate Health (Other); Corewell Health East (Other); Columbia Park Medical Group (Other); Humboldt Del Norte Independent Practice Association (Unknown); Metropolitan Health (Unknown); Park Nicollet Clinic (Other); PeaceHealth Medical Group (Other); Sanford Clinic (Unknown); TriHealth Inc. (Other); University Hospitals Medical Practices (Unknown); Warren Clinic (Unknown); Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 03527-06-C
Record Dates: First submitted 2008-06-09; First posted 2008-08-29 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2013-08

CONDITIONS: Hypertension
Keywords: hypertension; diabetes; quality improvement; blood pressure
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Quality Improvement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: quality improvement — 3-phase quality improvement intervention

SUMMARY:
Twelve health organizations from around the US were selected to participate in a chart review Hypertension and Diabetes Initiative with the goal of improving blood pressure control in persons with diabetes.

Hypothesis:

A three-phase quality improvement initiative facilitated and monitored through the International Diabetes Center (IDC) will result in improved population-mean systolic blood pressure in the aggregate data pool of patients from all 12 participating sites at geographically distinct health systems.

DETAILED DESCRIPTION:
Phase 1 - Preparation: Each participating site begins to organize itself for the project. Baseline data will be collected and will be used to benchmark where each site is relative to blood pressure control/management of persons with diabetes prior to the implementation of the training programs.

Phase 2 - Implementation: Sites begin to address the gaps they have identified that affect blood pressure outcomes of patients with diabetes. IDC provides two on-site training programs for providers and support staff.

Phase 3 - Follow-up: IDC provides on-going support to each site via individual and collaborative conference calls and resources on the project Web site. Patient and visit data (audit form) will be collected six and 12 months after training. This data will be compared to the site's pre-training data.

ELIGIBILITY:
Inclusion Criteria:

* ICD-9 Code 250 (indicates type 1 or type 2 diabetes)
* ICD- Code 648.0 (indicates pregnancy with type 1 or type 2 diabetes)
* ICD-9 Code 357.2 or 362.0, indicating complications of diabetes.
* A prescription for insulin or oral hypoglycemic agents
* Include those 18-75 years

Exclusion Criteria:

* Attend a dialysis unit (if the nephrologist is primary care manager)
* Have gestational diabetes (ICD-9 Code 648.8)
* Have a terminal illness (e.g., hospice patient)
* Do not have a documented blood pressure within the past year (this is asked on the audit form)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 11510 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 1 year

SECONDARY OUTCOMES:
Measure changes in action taken related to improving blood pressure management as percent of providers reporting changing (initiating or adjusting) blood pressure medication | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Powers, PhD, Principal Investigator — International Diabetes Center - Park Nicollet Institute; Robert M Cuddihy, MD, Principal Investigator — International Diabetes Center - Park Nicollet Institute

REFERENCES:
- [Background] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group; Lachin JM, Genuth S, Cleary P, Davis MD, Nathan DM. Retinopathy and nephropathy in patients with type 1 diabetes four years after a trial of intensive therapy. N Engl J Med. 2000 Feb 10;342(6):381-9. doi: 10.1056/NEJM200002103420603. PMID 10666428
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Saaddine JB, Cadwell B, Gregg EW, Engelgau MM, Vinicor F, Imperatore G, Narayan KM. Improvements in diabetes processes of care and intermediate outcomes: United States, 1988-2002. Ann Intern Med. 2006 Apr 4;144(7):465-74. doi: 10.7326/0003-4819-144-7-200604040-00005. PMID 16585660
- [Background] Adler AI, Stratton IM, Neil HA, Yudkin JS, Matthews DR, Cull CA, Wright AD, Turner RC, Holman RR. Association of systolic blood pressure with macrovascular and microvascular complications of type 2 diabetes (UKPDS 36): prospective observational study. BMJ. 2000 Aug 12;321(7258):412-9. doi: 10.1136/bmj.321.7258.412. PMID 10938049
- [Background] Major cardiovascular events in hypertensive patients randomized to doxazosin vs chlorthalidone: the antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT). ALLHAT Collaborative Research Group. JAMA. 2000 Apr 19;283(15):1967-75. PMID 10789664